CLINICAL TRIAL: NCT00993252
Title: Evaluation of an Active Strategy to Implement the Canadian CT Head Rule: Phase III
Brief Title: Canadian Computed Tomography (CT) Head Rule Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Ian Stiell, OHRI
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 42521; 2003165-01H
Record Dates: First submitted 2008-04-21; First posted 2009-10-12 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Head Injury
Keywords: head injury; radiography; clinical impact; dissemination
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: CT Scan — CT scan

SUMMARY:
Each year, Canadian emergency department physicians treat 600,000 patients with head injury. Many of these are adults with "minor head injury", i.e. loss of consciousness or amnesia and a Glasgow Coma Scale (GCS) score of 13-15. Only 6.2% of these "minor" patients have some acute injury on computed tomography (CT scan) and only 0.5% have an epidural hematoma requiring surgery. Among Canadian teaching hospital emergency departments, we have shown a fourfold variation in use of CT and that a small but important number of intracranial hematomas are missed at the first visit.

DETAILED DESCRIPTION:
Background: Each year, Canadian emergency department physicians treat 600,000 patients with head injury. Many of these are adults with "minor head injury", i.e. loss of consciousness or amnesia and a Glasgow Coma Scale (GCS) score of 13-15. Only 6.2% of these "minor" patients have some acute injury on computed tomography (CT scan) and only 0.5% have an epidural hematoma requiring surgery. Among Canadian teaching hospital emergency departments, we have shown a fourfold variation in use of CT and that a small but important number of intracranial hematomas are missed at the first visit. This renewal application builds on previous MRC/CIHR Health Services Research Committee funded grants to determine feasibility (phase 0, MRC GR-13304D, 1995-96), develop a clinical decision rule for CT in minor head injury (phase I, MRC MT-13700, 1996-99, N=3,121), and prospectively validate this Canadian CT Head Rule (phase II, CIHR #42521, 2000-03, N=2,707), all part of the U of Ottawa Group Grant in Decision Support Techniques (CIHR 2000-143). The Canadian CT Head Rule is comprised of simple clinical variables and allows physicians to be much more accurate in their diagnosis of brain injury and will standardize the use of CT without jeopardizing patient care (The Lancet 2001). In the recently completed prospective validation (phase II), we confirmed the accuracy and reliability of the rule in 2,707 additional patients.

Objectives: The goal of phase III is to evaluate the effectiveness and safety of an active strategy to implement the Canadian CT Head Rule into physician practice. Specific objectives are to: 1) Determine clinical impact by comparing the intervention and control sites for: a) CT Head ordering rates, b) Missed neurological intervention cases, c) Missed brain injuries, d) Number of deaths, d) Length of stay in ED, and e) Patient satisfaction; 2) Determine sustainability of the impact; 3) Evaluate performance of the Canadian CT Head Rule, with regards to: a) Accuracy, b) Physician accuracy in interpretation, and c) Physician comfort and compliance with use; 4) Conduct an economic evaluation to determine the potential for cost savings with widespread implementation; 5) Conduct an exploratory psychological process evaluation to examine whether physicians' intentions and behaviours can be predicted.

Methods: We propose a matched-pair cluster design study which compares outcomes during 3 consecutive 12-month 'before', 'after', and 'decay' periods at 6 pairs of 'intervention' and 'control' sites. These 12 hospital ED sites will be stratified as 'teaching' or 'community' hospitals, matched according to baseline CT head ordering rates, and then allocated within each pair to either intervention or control groups. During the 'after' period at the intervention sites, simple and inexpensive strategies will be employed to actively implement the Canadian CT Head Rule: a) physician group discussion and consensus, b) educational initiatives (lecture, posters, pocket cards), and c) a process-of-care modification with a mandatory reminder of the Rule at the point of requisition for radiography. These outcomes will be assessed: 1) Measures of clinical impact will compare the changes from 'before' to 'after' between the intervention and control sites: a) CT Head ordering proportions (the primary analysis); b) Number of missed brain injuries; c) Number of serious adverse outcomes; d) Length of stay in ED; e) Patient satisfaction. 2) Performance of the Canadian CT Head Rule: a) Accuracy of the rule; b) Physician accuracy of interpretation; c) Physician comfort and compliance. 3) Economic evaluation measures: a) CT head rate after discharge; b) Length of stay in ED and hospital; c) Hospital admission; d) Neurological intervention; e) Number of transfers. 4) Psychological Process Evaluation: Mail surveys of physicians before and after the intervention. During the 12-month 'decay' period, implementation strategies will continue, allowing us to evaluate the sustainability of the effect. We estimate a sample size of 2,400 patients in each period in order to have adequate power to evaluate the main outcomes.

Importance: This implementation study (phase III) is an essential step in the process of developing a new clinical decision rule / guideline for health care practitioners. Phase I successfully derived the Canadian CT Head Rule and phase II confirmed the accuracy and safety of the rule and, hence, the potential for physicians to improve care. What remains unknown is the actual change in clinical behaviour that can be effected by implementation of the Canadian CT Head Rule and whether implementation can be achieved with simple and inexpensive measures. We believe that the Canadian CT Head Rule has the potential to significantly limit health care costs and improve the efficiency of patient flow in busy Canadian EDs.

ELIGIBILITY:
Inclusion Criteria:

Consecutive adult patients presenting to one of the study hospital EDs after sustaining acute minor head injury will be enrolled into the study. Eligibility as an 'acute minor head injury' case will be determined by the patient having all of the following characteristics upon arrival in the ED.

1. Blunt trauma to the head resulting in witnessed loss of consciousness, definite amnesia, or witnessed disorientation, no matter how brief; this may be determined from the patient or from the report of a witness (the patient will be asked specific questions: 'do you remember the accident?', 'how did you get to the hospital?', 'have you talked to me before?').
2. Initial ED GCS score of 13 or greater as ascertained by the attending physician (e.g. opens eyes spontaneously, obeys commands, but speech may include only comprehensible but inappropriate words).
3. Injury within the past 24 hours.

Exclusion Criteria:

1. less than 16 years,
2. 'minimal' head injury i.e. no loss of consciousness, amnesia, or disorientation,
3. no clear history of trauma as the primary event (for example primary seizure or syncope),
4. GCS score of less than 13,
5. head injury occurred more than 24 hours previously,
6. obvious penetrating skull injury or depressed fracture,
7. acute focal neurological deficit (motor or cranial nerve) that cannot be ascribed to an extracerebral cause, for example, traumatic mydriasis or peripheral neuropathy,
8. have suffered a seizure prior to assessment in the ED,
9. a bleeding disorder or current use of oral anticoagulants,125 or
10. returned for reassessment of the same head injury

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4531 (Actual)
Dates: Start 2003-09; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Computed tomography ordering proportions | January 2009

SECONDARY OUTCOMES:
Number of missed CTs | January 2009
Number of serious adverse outcomes | January 2009
Length of stay in emergency department (ED) | January 2009
Patient satisfaction | January 2009
Sustainability of the intervention | January 2009
Performance of the Canadian CT Head Rule | January 2009
Economic evaluation measures | January 2009

CONTACTS AND LOCATIONS:
Overall Officials: Ian G Stiell, MD MSc, Principal Investigator — University of Ottawa
Locations (10):
- Canada (10):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Royal Columbian Hospital, Westminster, British Columbia
  - St. Thomas Hospital, Elgin, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Civic Campus, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook and Women's College HSC, Toronto, Ontario
  - Credit Valley Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Stiell IG, Clement CM, Grimshaw JM, Brison RJ, Rowe BH, Lee JS, Shah A, Brehaut J, Holroyd BR, Schull MJ, McKnight RD, Eisenhauer MA, Dreyer J, Letovsky E, Rutledge T, Macphail I, Ross S, Perry JJ, Ip U, Lesiuk H, Bennett C, Wells GA. A prospective cluster-randomized trial to implement the Canadian CT Head Rule in emergency departments. CMAJ. 2010 Oct 5;182(14):1527-32. doi: 10.1503/cmaj.091974. Epub 2010 Aug 23. PMID 20732978